CLINICAL TRIAL: NCT04266184
Title: Gebeliğe Bağlı Pelvik Kuşak Ağrısında Pelvik Kemer ve Kinezyo Bant Uygulamalarının Ağrı ve Fonksiyonel Mobilite Üzerine Etkileri
Brief Title: Effects of Pelvic Belt and Kinesio Tape on Pain and Functional Mobility in Pregnancy-Related Pelvic Girdle Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Muğla Sıtkı Koçman University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, İlkim Çıtak Karakaya, PT. PhD. Prof., Prof., Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 47921137-050.01.04-E.144981
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Pelvic Girdle Pain
Keywords: kinesio tape; pelvic belt; functional mobility; pain; kinesiophobia; neuroscience education; ergonomic education; activity limitation
MeSH Terms: conditions — Pelvic Girdle Pain; Pain; Kinesiophobia | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio tape (KT) (Experimental): Abdominal and symphisis pubis supported lumbopelvic KT will be applied. This group will also receive the same educational program with the control group.
  Interventions: Other: Kinesio tape (KT); Other: Educational program
- Pelvic belt (PB) (Active Comparator): A narrow and flexible adjustable pelvic belt will be used in high position (just under the spina iliaca anterior superior). This group will also receive the same educational program with the control group.
  Interventions: Other: Pelvic belt (PB); Other: Educational program
- Control group (Other): This group will receive a 1-hour educational program composed of neuroscience education and ergonomic training.
  Interventions: Other: Educational program

INTERVENTIONS:
Other: Kinesio tape (KT) — For abdominal taping, four I-shaped tapes will be used. Two of them will start from the superior symphisis pubis, follow the rectus abdominis muscle, and finish at the xiphoid process. Other two I-shaped tapes will start from the mid-symphisis pubis, follow the external oblique abdominals, and finish at the spina iliaca anterior superiors.
  Symphisis pubis taping will be applied with two I-shaped tapes, by forming a "X" shape.
  For lumbopelvic taping, three I-shaped KTs will be used. Two tapes will be applied bilaterally and longitudinally on the lumbar erector spinal muscles. The third tape will start from one sacroiliac joint and end at the other, vertically to the previous two tapes, forming a H-shape.
  All tapings will be applied with 15-25% tension (tape-off tension). KTs will stay three days. They will be removed from the site, and the skin will be checked and cleaned. Then, they will be reapplied for the next three days.
  Other Names: athletic tape; kinesiology tape; k tape; elastic tape
  Arms: Kinesio tape (KT)
Other: Pelvic belt (PB) — The women in this group will use the belts, after adjusting them at a comfortable tension, after getting up the bed in the mornings, during daily activities and walking. Evaluation will be made three days after the first application and they will be asked to continue using it for the second three-day period.
  Other Names: pelvic compression belt; maternity belt; sacroiliac support belt
  Arms: Pelvic belt (PB)
Other: Educational program — This program will include pain neuroscience education and ergonomic education, and will approximately last one hour.

SUMMARY:
This study investigates the effects of pelvic belt (PB) and kinesio taping (KT) applications on pain and functional mobility in pregnancy-related pelvic girdle pain (PGP), in comparison with the control group that received only pain neuroscience education and ergonomic training.

DETAILED DESCRIPTION:
Although there is strong evidence in the literature that pelvic support belts reduce pain in pregnancy-related pelvic girdle pain, no study investigating its effect on functional mobility with performance-based measurement methods or investigating its effectiveness on kinesiophobia has been found. Studies investigating the efficacy of KT in pregnant women with PGP are few and many are methodologically weak studies, most of which do not contain randomization and control groups. Also, no study has been found in the literature, which compares the effectiveness of PB and KT in pregnant women with PGP. Therefore, the primary aim of this study is to examine the effects of PB and KT on pain and functional mobility in pregnant women with PGP in comparison with the control group, which is only given pain neuroscience education and ergonomic training. The secondary aims are to investigate the effects of these applications on kinesiophobia, activity limitation and sleep quality; and to compare the groups in regard to patient compliance and treatment satisfaction levels of the groups.

ELIGIBILITY:
Inclusion Criteria:

* being able to read and write in Turkish
* being in 2nd or 3rd trimester of pregnancy
* having PGP for more than one week
* signing the informed consent form for the study

Exclusion Criteria:

* visual, auditory or cognitive problems which may prevent participation to the study
* health problems other than pregnancy-related PGP (orthopedic, neurologic, cardiorespiratory, etc.) or trauma history, which may affect standing from sitting, walking or stair climbing activities
* any gynecological or urological problems which may mimic pregnancy related PGP
* any diagnosed pregnancy complications other than PGP (preeclampsy, hypertension, diabetes,placental/fetal anomaly, preterm labor, etc.)
* high risk pregnancy (multiple gestation, etc.)
* history of spinal injury, ankylosing spondilitis, rheumatoid arthritis, intervertebral disc pathology)
* A positive straight leg raise test result, as well as sensory or motor deficits indicating intervertebral disc pathology
* history of prepregnancy low back or pelvic girdle pain
* using any analgesic or myorelaxant medication
* contraindications to KT or PB (impaired skin integrity or lesion in the lumbopelvic and abdominal regions, history of allergic reaction, etc.)
* previous KT (abdominal or lumbosacral) or PB experience

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
change in general pain intensity during activity | baseline, approximately one-hour after the first intervention, three days after the first intervention, one week after the first intervention, and one week after cessation of intervention
  The women will be asked to mark their pain intensity during activities in general. 0 (no pain)-10 cm (unbearable pain) visual analogue scale will be used.
change in pain intensity during five times sit to stand test | baseline, approximately one-hour after the first intervention, three days after the first intervention, one week after the first intervention, and one week after cessation of intervention
  The women will be asked to mark their pain intensity during five times sit to stand test. 0 (no pain)-10 cm (unbearable pain) visual analogue scale will be used.
change in pain intensity during five-stairs climbing test | baseline, approximately one-hour after the first intervention, three days after the first intervention, one week after the first intervention, and one week after cessation of intervention
  The women will be asked to mark their pain intensity during five-stairs climbing test. 0 (no pain)-10 cm (unbearable pain) visual analogue scale will be used.
change in pain intensity during timed up and go test | baseline, approximately one-hour after the first intervention, three days after the first intervention, one week after the first intervention, and one week after cessation of intervention
  The women will be asked to mark their pain intensity during timed up and go test. 0 (no pain)-10 cm (unbearable pain) visual analogue scale will be used.
change in impairment during active straight leg raise test | baseline, approximately one-hour after the first intervention, three days after the first intervention, one week after the first intervention, and one week after cessation of intervention
  The women will be asked to score their impairment during active straight leg raise test. 0 (not difficult at all)-5 (unable to do) scoring system will be used. Scores for right and left legs will be summed and recorded.

SECONDARY OUTCOMES:
change in kinesiophobia | baseline, three days after the first intervention, one week after the first intervention, and one week after cessation of intervention
  Turkish version of Tampa Kinesiophobia Scale will be used. The score ranges between 17 and 68, and higher score indicates higher kinesiophobia.
change in activity limitation | baseline, three days after the first intervention, one week after the first intervention, and one week after cessation of intervention
  Turkish version of Pelvic Girdle Questionnaire will be used. Total score varies between 0 and 75, and higher score indicates higher activity limitation.
change in sleep quality | baseline, three days after the first intervention, one week after the first intervention, and one week after cessation of intervention
  Quality of sleep will be assessed on a 0 (very bad)-10 (very good) cm VAS.
patient compliance | baseline, three days after the first intervention, one week after the first intervention, and one week after cessation of intervention
  For PB and KT groups, comfort and easiness of using PB and KT will be assessed by 0 (not at all)-10 (extremely comfortable/easy) cm VASs. All groups will be questioned about the comprehensibility of the educational program on 0 (not at all)-10 (completely comprehensible) cm VASs. Also, degree of following the suggestions given in the educational program will be evaluated by 0 (not at all)-10 (completely) cm VASs.
treatment satisfaction | baseline, three days after the first intervention, one week after the first intervention, and one week after cessation of intervention
  Treatment satisfaction will be assessed by 0 (not at all)-10 (extremely satisfactory) cm VASs.

CONTACTS AND LOCATIONS:
Overall Officials: İlkim Çıtak Karakaya, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Bodes Pardo G, Lluch Girbes E, Roussel NA, Gallego Izquierdo T, Jimenez Penick V, Pecos Martin D. Pain Neurophysiology Education and Therapeutic Exercise for Patients With Chronic Low Back Pain: A Single-Blind Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Feb;99(2):338-347. doi: 10.1016/j.apmr.2017.10.016. Epub 2017 Nov 11. PMID 29138049
- [Background] Draper C, Azad A, Littlewood D, Morgan C, Barker L, Weis CA. Taping protocol for two presentations of pregnancy-related back pain: a case series. J Can Chiropr Assoc. 2019 Aug;63(2):111-118. PMID 31564749
- [Background] Bertuit J, Van Lint CE, Rooze M, Feipel V. Pregnancy and pelvic girdle pain: Analysis of pelvic belt on pain. J Clin Nurs. 2018 Jan;27(1-2):e129-e137. doi: 10.1111/jocn.13888. Epub 2017 Nov 3. PMID 28544276